CLINICAL TRIAL: NCT00826085
Title: A Phase I/II Study Evaluating the Maximum Tolerated Dose, Bioequivalence/Pharmacokinetics, Safety, and Efficacy of Hyperthermia and ThermoDox (Lyso-Thermosensitive Liposomal Doxorubucin) in Patients With Local-Regional Recurrent Breast Cancer.
Brief Title: Phase 1/2 Study of ThermoDox With Approved Hyperthermia in Treatment of Breast Cancer Recurrence at the Chest Wall
Acronym: DIGNITY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imunon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105-08-201
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Recurrent Chest Wall Cancer; Loco-regional Recurrent Breast Cancer; Breast Cancer Recurrence at the Chest Wall
MeSH Terms: conditions — Breast Neoplasms | interventions — Hot Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thermodox in combination with hyperthermia (Experimental): Single arm study
  Interventions: Drug: ThermoDox in combination with Microwave Hyperthermia (heat)

INTERVENTIONS:
Drug: ThermoDox in combination with Microwave Hyperthermia (heat) — ThermoDox is a 30 minute intravenous infusion followed by hyperthermia within 60 minutes of infusion completion.
  Hyperthermia is a therapy used to heat tumors for 60 minutes. Using heat energy, the tumor is heated to a certain temperature. The heat can damage cancer cells at levels that are usually safe for normal cells and can be used to attack cancer in four major ways: 1) heat damages or weakens the cells of the tumor; 2) heat increase blood flow through the weakened tumor; 3) increased blood flow raises oxygen levels in tumors; and 4) when the body senses fever it can stimulate the nature immune system.
  All patients will receive up to six ThermoDox/hyperthermia treatments at 21-day intervals.

SUMMARY:
This is a research study to evaluate the effects of ThermoDox in combination with therapeutic heating of the chest wall in the treatment of recurrent regional breast cancer. The purpose of this study is to evaluate the bioequivalence of ThermoDox and measure efficacy in recurrent chest wall patients.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women in both the United States and the world. Despite a variety of hormonal, cytotoxic and biologic approaches, a significant number of tumors will recur in the chest wall and axillary area following primary treatment. Any local recurrence of breast cancer after mastectomy is generally regarded as a poor prognostic indicator. However, it is also generally agreed that those who present without measurable metastatic disease at the time of loco-regional recurrence (LRR) have a more favorable disease and may experience long-term survival. Overall up to 35% of women with operable breast cancer will experience an isolated LRR following their primary treatment. Patients with LRR suffer from disfiguring tumors and other clinical signs and symptoms including pain, lymphedema limiting range of motion in the affected extremity, foul-smelling wounds, and a visual reminder of tumor progression. Up to 40% of patients undergoing a mastectomy as their primary treatment will experience a recurrence at the chest wall or overlying skin (RCW).

For initial curative intent in LRR, available interventions include surgical resection in patients whose tumor and clinical status permits anesthesia and surgical removal, radiation therapy in patients whose tumor and clinical status permits additional radiation, systemic hormonal and/or cytotoxic chemotherapy in patients whose tumors are sensitive to such drugs and combinations of the aforementioned. For unresectable LRR tumors, radiation and chemotherapy are used to manage the disease. In this setting some success has been achieved; however, a patient who reoccurs following these treatments is often treated with palliative intent.

Diathermy refers to the therapeutic generation of local heat in body tissues by high-frequency electromagnetic radiation, electric currents, or ultrasonic waves. In mild hyperthermia local tissue temperatures are restricted to a range of 39-45°C. Two types of external devices, microwave systems and ultrasound systems, have been approved by the FDA for delivering mild hyperthermia to the chest wall.

Mild hyperthermia from either microwave or ultrasound devices has been used safely in breast cancer treatment. In conjunction with external beam radiation, both types of devices have been used to heat the chest wall and both devices have demonstrated enhanced effects when compared to radiation therapy without additional hyperthermia.

Doxorubicin hydrochloride is a cytotoxic anthracycline antibiotic. The recommended single-agent dose of doxorubicin HCl (Adriamycin®) for injection is 60 to 75 mg/m2 intravenously (IV) in three-week cycles. Acute myelosuppression and long term, cumulative, cardiotoxicity (congestive heart failure) are dose-limiting. Doxorubicin is active against breast cancer as a single agent and is used with other drugs in multi-agent chemotherapy regimens. In LRR breast cancer, single agent doxorubicin achieves response rates comparable to combination chemotherapy.

Lyso-thermosensitive liposomal doxorubicin (ThermoDox®) is a temperature sensitive liposomal drug delivery system that selectively accumulates in tumors as a result of their leaky vasculature. During ThermoDox/hyperthermia therapy, the tumor is heated locally while the rest of the body remains at a normal temperature. When the liposomes encounter a temperature of 39.5°C or above, they release doxorubicin locally into the heated area. Liposomal doxorubicin is administered intravenously and, because it is particulate, will eventually be removed from circulation by the reticuloendothelial system in the liver and spleen. Pharmacokinetic data from liver cancer patients treated with radiofrequency ablation (RFA) and ThermoDox show that the major portion of exposure to ThermoDox (about 95% of the liposomal doxorubicin plasma AUC0-∞) occurs during the first six hours following the infusion, establishing this time period as optimal for application of hyperthermia. Animal studies have repeatedly shown higher tumor doxorubicin concentrations and enhanced tumor cell killing when ThermoDox is combined with hyperthermia compared to doxorubicin without hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented recurrent/metastatic adenocarcinoma of the breast with a recurrence on the chest wall (or its overlying skin):

   * Subjects with ulcerative chest wall disease defined as non-healing wounds consistent with cancer are eligible.
   * Subjects with prior skin changes consistent with inflammatory breast carcinoma are eligible.
   * Breast carcinoma for medical reasons not being resected
2. Tumor thickness must be clinically indicated for hyperthermia therapy, as measured by clinical exam or imaging studies (CT or MRI). The target local tumor lesion(s) must be able to be covered within two hyperthermia fields of treatment.
3. Disease that has progressed despite other available standard treatment options, based on what is clinically indicated according to the investigator's clinical and medical judgment, including:

   * One or more radiation treatment(s) to the chest wall or breast up to a maximum prior dose of 12,000 cGy in the hyperthermia field (not administered less than 28 days prior to enrollment).
4. Subjects who have previously received hyperthermia in conjunction with either radiation therapy or chemotherapy are eligible.
5. Subjects may have distant metastasis, including brain metastases. Subjects with known brain metastases are eligible if:

   * They have received standard anti-tumor treatment for their brain metastases without encephalopathy;
   * Their neurological function is stable for at least 30 days and either off steroid therapy or on a stable steroid regimen.
6. Non-pregnant female at least 18 years of age. If the subject is of child-bearing age, must have a negative serum pregnancy test at baseline and must agree to practice an acceptable form of birth control while on the study.
7. Provide written informed consent and willing to comply with protocol requirements.

Exclusion Criteria:

1. Requires any concomitant antineoplastic therapy. Prior chemotherapy should not be administered within 5 half-lives or 28 days whichever is shorter. Subjects on a current stable dose of hormonal treatments may continue on a stable dose during the study (i.e. arimidex, amarosin, herceptin).
2. Prior confirmed allergic reaction (including moderate rash, dyspnea, wheezing, urticaria or other symptoms) attributed to the administration of either anthracyclines or other liposomally encapsulated drugs that required discontinuation of prior therapy.
3. Prior therapy with anthracyclines exceeding the following doses (subjects will be discontinued at 600 mg/m2 lifetime dose irrespective of the number of ThermoDox® cycles received):

   Free (i.e., non-liposomal) or liposomal doxorubicin > 450 mg/m2 Free epirubicin > 900 mg/m2.
4. Previous (required active treatment within 5 years) or concomitant malignancy except basal cell cancer, in situ carcinoma of the cervix, or contralateral breast cancer. Subjects with a prior contralateral breast malignancy can be included if they did not receive any chemotherapy.
5. Baseline laboratories (repeat labs can be evaluated at baseline to establish eligibility):

   * ANC Granulocytes < 1,500/ microliter
   * Platelets < 75,000/ microliter
   * Hemoglobin < 9 gm/dL
   * Total Bilirubin > 2 mg/dL
   * ALT and AST > 2.5 X upper limit of normal
   * Creatinine > 1.5 X upper limit of normal.
6. ECOG/Zubrod Performance Status > 2.
7. MUGA/Echocardiogram Left Ventricular Ejection Fraction < 50%.
8. Has a medical or psychiatric condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations.
9. History of:

   * Acute coronary syndrome
   * Cerebral vascular accident
   * Abnormal cardiac stress testing within last 6 months
   * Symptomatic coronary artery disease
   * Uncontrolled hypertension or cardiomyopathy
   * Cardiac valvular surgery or open heart surgery
   * Known structural heart disease.
10. Has a condition which may interfere with the hyperthermia portion of the trial such as: functioning cardiac pacemaker; metal plates, rods or prosthesis of the chest wall, breast reconstruction with implants, severe numbness and/or tingling of the chest wall or breast, skin grafts and/or flaps on the breast or chest wall.
11. Active infection requiring antibiotic treatment
12. Has received any external radiation therapy within 28 days prior to enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To determine the bioequivalence of ThermoDox when used with hyperthermia among patients with RCW breast cancer. | PK collection at Cycle 1 and Cycle 2
To determine efficacy of ThermoDox in combination with Hyperthermia | Efficacy assessed at Cycle 3, Cycle 5 and End of Treatment

SECONDARY OUTCOMES:
To evaluate the safety of ThermoDox in combination with Hyperthermia | Through 6 treatment Cycles

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Borys, MD, Study Director — Imunon
Locations (6):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - Southeastern Regional Medical Center, Newnan, Georgia
  - University of Maryland, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Southwestern Regional Medical Center, Tulsa, Oklahoma
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Zagar TM, Vujaskovic Z, Formenti S, Rugo H, Muggia F, O'Connor B, Myerson R, Stauffer P, Hsu IC, Diederich C, Straube W, Boss MK, Boico A, Craciunescu O, Maccarini P, Needham D, Borys N, Blackwell KL, Dewhirst MW. Two phase I dose-escalation/pharmacokinetics studies of low temperature liposomal doxorubicin (LTLD) and mild local hyperthermia in heavily pretreated patients with local regionally recurrent breast cancer. Int J Hyperthermia. 2014 Aug;30(5):285-94. doi: 10.3109/02656736.2014.936049. PMID 25144817